CLINICAL TRIAL: NCT07321587
Title: Activity Tracking, Care Partner Co-participation, Text Reminders, Instructional Education, Video-Guided Physical Rehabilitation, and Exercise (ACTIVE) Intervention Among Older Adults With and Without Mild Dementia
Brief Title: Activity Tracking, Care Partner Co-participation, Text Reminders, Instructional Education, Video-Guided Physical Rehabilitation, and Exercise
Acronym: ACTIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 25-01158
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Mild Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention, then Control (Experimental): Week 1 (Pre-Intervention): Participants will wear the Fitbit smartwatch during waking hours. Data collected during this week will serve as baseline and for troubleshooting technical issues.
  Weeks 2-4 (Intervention): Participants will receive the ACTIVE intervention (Activity tracking, Care partner co-participation, Text reminders, Instructional education, Virtual physical therapy and Exercise).
  Week 5 (Crossover/Washout): Participants will switch arms (intervention to control).
  Weeks 6-8 (Control): Participants will continue in the control arm (Fitbit use only).
  Interventions: Behavioral: ACTIVE Intervention
- Control, then Intervention (Experimental): Week 1 (Pre-Control): Participants will wear the Fitbit smartwatch during waking hours. Data collected during this week will serve as baseline and for troubleshooting technical issues.
  Weeks 2-4 (Control): Participants will continue in the control arm (Fitbit use only).
  Week 5 (Crossover/Washout): Participants will switch arms (control to intervention).
  Weeks 6-8 (Intervention): Participants will the ACTIVE intervention (Activity tracking, Care partner co-participation, Text reminders, Instructional education, Virtual physical therapy and Exercise).
  Interventions: Behavioral: ACTIVE Intervention

INTERVENTIONS:
Behavioral: ACTIVE Intervention — The ACTIVE Intervention comprises the following components:
  * Fitbit Smartwatch-Based Activity Tracking
  * Care Partner Co-Participation
  * Motivational Text Messaging
  * Instructional Education Videos
  * Virtual Physical Therapy
  * Exercise (Walking Exercise)

SUMMARY:
This is a multi-methods two-arm, crossover, analyst-blinded randomized controlled trial with embedded qualitative interviews, enrolling 50 dyads (older adult-care partner). Participants will receive the ACTIVE intervention, which includes a Fitbit smartwatch, motivational text messages to engage in walking exercise, instructional educational videos, and virtual physical therapy sessions. Intervention components will be delivered over 3 weeks, with continuous monitoring of physical activity via Fitbit data, read receipts of the motivational text messages, and log of engagement in the virtual physical therapy and educational videos.

ELIGIBILITY:
Inclusion Criteria:

Older Adults:

* Age ≥65 years.
* With or without mild dementia.
* Willing to consent to participate in the study or have an LAR that is willing to consent for their participation in the study
* Willing to wear a Fitbit smartwatch, receive text messages, watch intervention-related videos, participate in physical therapy, and walking exercise.
* No contraindications to engaging in physical activity.

Care Partners:

* Age ≥18 years.
* Met criteria for survey participation.
* Person being cared for is recruited in the study.
* Willing to consent to participation
* Willing to wear a Fitbit smartwatch, receive text messages, watch intervention-related videos, participate in physical therapy, and walking exercise.
* No contraindications to engaging in physical activity.

Exclusion Criteria:

Older Adults:

* Severe cardiac, neurologic, or musculoskeletal condition (including but not limited to recent or untreated fracture in any part of the body)
* limiting participation in daily walking or Fitbit smartwatch use.
* Moderate to severe dementia (using the clinical dementia rating scale of 2 or higher
* Inability to operate or manage a Fitbit smartwatch device (even with care partner support).
* No phone or phone not capable of receiving text messages or watching videos.
* No internet for watching videos

Care Partners:

* Severe cardiac, neurologic, or musculoskeletal condition limiting participation in daily walking or Fitbit smartwatch use.
* Pregnant care partners
* Any level of dementia or cognitive impairment among care partners
* Inability to operate or manage a Fitbit smartwatch device.
* Inability to co-participate in intervention tasks with older adult
* No phone or phone not capable of receiving text messages or watching videos.
* No internet for watching videos

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adoption | Up to Week 7 (End of Week 1 of Intervention Period)
  Measured as the proportion of participants who initiate use of each intervention component:
  * Smartwatch: device activated and worn for ≥3 days during week 1.
  * Text reminders: ≥1 responses to text message opened/read in week 1.
  * Virtual PT videos: at least one session accessed in week 1, which will be tracked online through participant specific username.
  * Instructional education videos: at least one video accessed in week 1,which will be tracked online through participant specific username.
Feasibility: Smartwatch | Up to Week 8
  Measured as sustained engagement with each component during the 3-week intervention:
  * Smartwatch: proportion of days with ≥8 hours of wear time (captured on Fitabase).
    * Text reminders: proportion of responses to text messages (captured on Fitabase) opened or acknowledged.
    * Virtual PT videos: proportion of assigned sessions completed (captured on myACTIVEsteps.com via username); feasibility target.
    * Instructional education videos: proportion of assigned videos completed (captured on myACTIVEsteps.com via username.
Feasibility: Motivational Texts | Up to Week 8
  Measured as sustained engagement with each component during the 3-week intervention:
  * Text reminders: proportion of responses to text messages (captured on Fitabase) opened or acknowledged.
    * Virtual PT videos: proportion of assigned sessions completed (captured on myACTIVEsteps.com via username); feasibility target.
    * Instructional education videos: proportion of assigned videos completed (captured on myACTIVEsteps.com via username.
Feasibility: Virtual Physical Therapy | Up to Week 8
  Measured as sustained engagement with each component during the 3-week intervention:
  * Virtual PT videos: proportion of assigned sessions completed (captured on myACTIVEsteps.com via username); feasibility target.
    * Instructional education videos: proportion of assigned videos completed (captured on myACTIVEsteps.com via username.
Feasibility: Instructional Education Videos | Up to Week 8
  Measured as sustained engagement with each component during the 3-week intervention:
  * Instructional education videos: proportion of assigned videos completed (captured on myACTIVEsteps.com via username.
Acceptability: System Usability Scale (SUS) | Up to Week 10
  The SUS is a 10-item survey assessing the usability of a system. Each item is rated on a Likert scale from 1-5; the raw score is the sum of responses, which is transformed to a standardized score ranging from 0-100; higher scores indicate greater usability.
Acceptability: Perceived Usefulness (PU): Smartwatch | Up to Week 10
  The PU survey is a 5-item assessment of perceived usefulness of technology. Each item is rated on a Likert scale from 1-7. The score is calculated as the average of responses and ranges from 1-7; higher scores indicate greater perceived usefulness.
Acceptability: Perceived Usefulness (PU): Motivational Texts | Up to Week 10
  The PU survey is a 5-item assessment of perceived usefulness of technology. Each item is rated on a Likert scale from 1-7. The score is calculated as the average of responses and ranges from 1-7; higher scores indicate greater perceived usefulness.
Acceptability: Perceived Usefulness (PU): Instructional Education Videos | Up to Week 10
  The PU survey is a 5-item assessment of perceived usefulness of technology. Each item is rated on a Likert scale from 1-7. The score is calculated as the average of responses and ranges from 1-7; higher scores indicate greater perceived usefulness.
Acceptability: Perceived Usefulness (PU): Virtual Physical Therapy | Up to Week 10
  The PU survey is a 5-item assessment of perceived usefulness of technology. Each item is rated on a Likert scale from 1-7. The score is calculated as the average of responses and ranges from 1-7; higher scores indicate greater perceived usefulness.
Acceptability: Perceived Ease-of-Use (PEU): Smartwatch | Up to Week 10
  The PEU survey is a 5-item assessment of perceived ease-of-use of technology. Each item is rated on a Likert scale from 1-7. The score is calculated as the average of responses and ranges from 1-7; higher scores indicate greater perceived ease-of-use.
Acceptability: Perceived Ease-of-Use (PEU): Motivational Texts | Up to Week 10
  The PEU survey is a 5-item assessment of perceived ease-of-use of technology. Each item is rated on a Likert scale from 1-7. The score is calculated as the average of responses and ranges from 1-7; higher scores indicate greater perceived ease-of-use.
Acceptability: Perceived Ease-of-Use (PEU): Instructional Education Videos | Up to Week 10
  The PEU survey is a 5-item assessment of perceived ease-of-use of technology. Each item is rated on a Likert scale from 1-7. The score is calculated as the average of responses and ranges from 1-7; higher scores indicate greater perceived ease-of-use.
Acceptability: Perceived Ease-of-Use (PEU): Virtual Physical Therapy | Up to Week 10
  The PEU survey is a 5-item assessment of perceived ease-of-use of technology. Each item is rated on a Likert scale from 1-7. The score is calculated as the average of responses and ranges from 1-7; higher scores indicate greater perceived ease-of-use.
Intervention Delivery Fidelity | Up to Week 8.
  Proportion of intervention components successfully delivered by study staff.
Participant Fidelity | Up to Week 8.
  Proportion of assigned intervention activities completed, verified via Fitbit logs, video analytics, and message tracking.
Change in Falls Efficacy Scale-International (FES-I) Score | Baseline, Up to Week 10
  FESI-I is a 16-item self-report questionnaire assessing older adults' fear about falling during daily activities. Each item is rated on a Likert scale from 1-4 (not at all to very concerned). The total score is the sum of responses and ranges from 16-64, where higher scores mean more fear and less confidence.
Change in Activities of Daily Living (ADL) Score | Baseline, Up to Week 10
  The ADL ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. Participants are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
Change in Instrumental Activities of Daily Living (IADL) Score | Baseline, Up to Week 10
  IADL is an 8-item assessment of independence in completing complex tasks. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women and 0 through 5 for men to avoid potential gender bias.
Change in Knowledge, Attitude, and Practice (KAP) of Physical Exercise: Knowledge Score | Baseline, Up to Week 10
  The Knowledge subsection of the KAP survey comprises 20 items assessing knowledge of physical exercise. Each item is rated on a Likert scale from 1-5. The total score is the sum of responses and ranges from 20-100; higher scores indicate greater knowledge.
Change in Knowledge, Attitude, and Practice (KAP) of Physical Exercise: Attitude Score | Baseline, Up to Week 10
  The Attitude subsection of the KAP survey comprises 10 items assessing attitude toward physical exercise. Each item is rated on a Likert scale from 1-5. The total score is the sum of responses and ranges from 10-50; higher scores indicate more positive attitude toward physical exercise.
Change in Knowledge, Attitude, and Practice (KAP) of Physical Exercise: Attitude Score | Baseline, Up to Week 10
  The Practice subsection of the KAP survey comprises 10 items assessing practice of physical exercise. Each item is rated on a Likert scale from 1-5. The total score is the sum of responses and ranges from 10-50; higher scores indicate greater practice of physical exercise.
Change in Short Form - 12 Quality of Life Survey (SF-12) | Baseline, Up to Week 10
  The SF-12 is a 12-item assessment of quality of life. Each item is rated on a Likert scale from 1-5. The raw score is the sum of responses; the raw score is converted to a standardized score ranging from 0-100 with a mean of 50 and standard deviation of 10. Higher scores indicate greater quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dowin Boatright, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Oluwaseun.Adeyemi@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Oluwaseun.Adeyemi@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.